CLINICAL TRIAL: NCT04378738
Title: The Role of Social Media as an Information Source in Covid19 Pandemic
Brief Title: Social Media and Covid19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AcibademU social media
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Social Media; Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: a survey study of a cohort about social media awareness regarding coronavirus pandemic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): the healthy people who accepted to participate in the study
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: survey — all people in the cohort

SUMMARY:
According to the data of February 2020, in Turkey with a population of 83.9 million, internet and social media usage percentage to population are 74% and 64% respectively. Although previous researches have investigated the effect of social media on different medical situations, there is no study focused role of social media on patients' behavior and information source during the COVID-19 pandemic. In the present study, it is aimed to reveal the impact of social media on patients' attitudes and information sources during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The coronavirus disease (COVID-19) outbreak was first diagnosed in late December 2019 in Wuhan at China's Hubei province. After four months, coronavirus infection has spread to 6 continents and 185 countries, with a dramatic increase of almost 3 million people have been infected and more than 200,000 people died.JHM As a result of the pandemic, the closure of borders, social isolation, and the crushing of health systems under an excessive load, peoples search different ways to achieve proper information regarding protecting themselves from this disaster including government announcements, hospitals, private doctors, and social media.

According to the data of February 2020, in Turkey with a population of 83.9 million, internet and social media usage percentage to population are 74% and 64% respectively. Social media is the most frequently translated way of informing due to its quick, cheap, and easy access potential.

Although previous researches have investigated the effect of social media on different medical situations, there is no study focused role of social media on patients' behavior and information source during the COVID-19 pandemic. In the present study, it is aimed to reveal the impact of social media on patients' attitudes and information sources during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 yo
* no diagnosis with any psychologic disease
* with literacy

Exclusion Criteria:

* younger than 18 yo
* inability to complete the form
* not giving consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-07 (Estimated); Study Completion 2020-05-08 (Estimated)

PRIMARY OUTCOMES:
the role of social media | 1 week
  applying a custom made survey to examine the role of social media and which type of research module is more effective

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bahar Yuksel, Istanbul
  - Haseki Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
if requested to.

REFERENCES:
- [Result] Khoong EC, Rivadeneira NA, Hiatt RA, Sarkar U. The Use of Technology for Communicating With Clinicians or Seeking Health Information in a Multilingual Urban Cohort: Cross-Sectional Survey. J Med Internet Res. 2020 Apr 6;22(4):e16951. doi: 10.2196/16951. PMID 32250280